CLINICAL TRIAL: NCT00588978
Title: Longitudinal Impact of Diet and/or Exercise-induced Weight Loss on Metabolic Markers of Cardiovascular Disease
Brief Title: Impact of Diet and/or Exercise-induced Weight Loss on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Barbara I Gulanski, MD, MPH, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25094
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases
Keywords: c-reactive protein; obesity; women's cardiovascular health
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Diet alone
  Interventions: Behavioral: diet and/or exercise
- 2 (Active Comparator): Exercise alone
  Interventions: Behavioral: diet and/or exercise
- 3 (Active Comparator): Diet and exercise (combined)
  Interventions: Behavioral: diet and/or exercise

INTERVENTIONS:
Behavioral: diet and/or exercise — Three arms are included: Diet Alone, Exercise Alone, and Combined Diet and Exercise

SUMMARY:
The purpose of this pilot study is to examine the effect of diet and/or exercise-induced weight loss on nontraditional cardiovascular risk factors such as c-reactive protein, insulin levels and sex steroids in obese postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* obese postmenopausal women
* able to exercise
* non-smokers

Exclusion Criteria:

* cardiovascular disease
* medications that would interfere with outcome measures (e.g., including ACE inhibitors, lipid lowering medications, beta-blockers, etc)
* known diabetes

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-08-01 (Actual); Primary Completion 2007-02-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
c-reactive protein | baseline, every 1-2 weeks during intervention , then end-of-study

SECONDARY OUTCOMES:
HOMA (measure of insulin resistance) and sex steroids | baseline, every 1-2 weeks during intervention, then end-of-study

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Gulanski, MD, MPH, Principal Investigator — Yale Univeristy School of Medicine
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States